CLINICAL TRIAL: NCT03873103
Title: The Belgian Molecular Profiling Program of Metastatic Cancer for Clinical Decision and Treatment Assignment - Precision 1
Brief Title: The Belgian Molecular Profiling Program of Metastatic Cancer for Clinical Decision and Treatment Assignment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Belgian Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: BSMO 2014-2
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PRECISION 1 will enroll patients with metastatic solid tumors. The local PI will verify if the candidate patient fits the inclusion/ exclusion criteria.

The participant will sign the PRECISION 1 informed consent. NGS data will be collected from local panel testing on DNA extracted from tissue samples or plasma.

Data will be collected from further molecular testing performed at the different laboratories: select rearrangements (fusion genes and translocations) by RT PCR, FISH or NGS; copy number variations of selected genes via the NGS platform (if possible) or using FISH or other technologies such as SNP arrays in case the NGS technology is incapable of giving this information.

Results will be stored in the Precision Belgium section of the Healthdata database.

Data on germline variants will also be collected in the Healthdata database whenever this information is available.

The cooperating clinical investigator will decide with the patient the treatment strategy, -guided by the best interest of the patient and the availability of respective options :

* " Empirical " available approved treatment (for example chemotherapy, immunotherapy)
* Genotype-driven standard of care
* Inclusion in a genotype-matched clinical trial (includes signing of trial-specific IC)
* Inclusion in PRECISION 2 if options 2/3 not available. Irrespective of treatment choice, the patient will be followed by the collaborating clinician and will have follow-up data collected every 6 months for determination of disease status and survival endpoints.

Clinical data will be collected and stored in the Healthdata database. Genomic data (somatic and germline whenever available) and clinical data (tumor type and stage, number of previous lines, treatment choice, response rate, PFS on chosen and previous treatments, …) will be uploaded on the Healthdata platform and can be consulted via password-protected web access by the local PI at each participating center. European regulation protecting patient privacy will apply ("GDPR").

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid tumors that are candidates for systemic therapy (early lines are preferred).
* Patient showing an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Patients able to provide written informed consent prior to enrollment into a subsequent clinical trial.
* Patients agrees to provide NGS data (somatic and/or germline) as well as clinical data baseline and during follow-up.

Exclusion Criteria:

* Life expectancy of less than 12 weeks.
* Inability to comply with protocol procedures.
* Known presence of severe hematopoietic, renal, and/or hepatic dysfunction (according to the local PI).
* Targeted gene sequencing on DNA extracted from decalcified bone biopsies is not accepted.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 patients with metastatic solid tumors that are eligible for systemic therapy will be recruited at 7 Belgian academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with "actionable" driven mutations. | 18 months
Percentage of patients enrolled in genomics-driven clinical trials and in the PRECISION 2 clinical trial. | 18 months
Clinical benefit rate as defined by survival and/or objective response rate and rate of stable disease lasting more than 6 months with genomics-driven therapy in non-approved indications | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Aftimos, Dr, Principal Investigator — Institute Jules Bordet
Locations (10):
- Belgium (10):
  - ZNA, Antwerp
  - GZA, Antwerp
  - AZ Klina, Brasschaat
  - Institute Jules Bordet, Brussels
  - AZ VUB, Brussels
  - Les Cliniques Universitaires St Luc, Brussels
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
  - CHU Sart-Tilman, Liège
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No